CLINICAL TRIAL: NCT03913208
Title: Priority to Cryopreservation Strategy (PCS) in IVF-ICSI Cycles is it Going to Make the Difference?
Brief Title: Priority to Cryopreservation Strategy (PCS) in IVF-ICSI Cycles
Acronym: PCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Infertility; IVF; ICSI; Cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Will be subjected to priority to freeze
  Interventions: Procedure: Priority to freeze
- Control group (Active Comparator): Will receive fresh embryo transfere
  Interventions: Procedure: Fresh embryo transfer

INTERVENTIONS:
Procedure: Priority to freeze — Priority for cryopreservation and later on embryo transfer in artificial cycle with endometrium preparation by the exogenous administration of estrogen-progesterone.
  Arms: Study group
Procedure: Fresh embryo transfer — usual strategy of giving the priority for fresh embryo transfer
  Arms: Control group

SUMMARY:
This multicentre randomized controlled trial will be done to evaluate a new strategy in IVF-ICSI practice that gives that priority to freeze for the embryos and goes to fresh embryo transfer only if at least one set of same quality embryos is available for cryopreservation.

DETAILED DESCRIPTION:
This study will be a non-blind, prospective, double-armed, randomized clinical trial. The study will be conducted at five centers, the Educational Hospital Fertility Unit of Tanta University, the fertility center of Cairo University, the fertility center of Assiut University, the Egyptian Consultants Fertility Center in Tanta, and MRC fertility center in Cairo from May 1st 2019 till the end of the objected number. The study will be conducted in accordance with the Declaration of Helsinki, and all participants should sign a written informed consent before inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for IVF/ICSI
* Presence of good number of embryos > 5

Exclusion Criteria:

* Low quality embryos
* Low ovarian reserve
* Low number of embryos

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative pregnancy rates | 3 months
  The number of pregnant women in both groups after 3 cycles

SECONDARY OUTCOMES:
Failure of pregnancy | 3 months
  Failed ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elhalwagy, MD, Study Director — Tanta Universit; Yaser Mesbah, MD, Study Chair — Mansiura University; Ahmed Abbas, MD, Study Chair — Assiut University; Ahmed Elsawaf, MD, Study Chair — Cairo University; Shereef Elshowaikh, MD, Study Chair — Tanta University; Abdelghaffar Dawood, MD, Study Chair — Tanta University; Ahmed Elkhyat, MD, Study Chair — Tanta University; Shereen Elbohoty, MD, Study Chair — Tanta University; Waleed Mamdouh, MD, Study Chair — Tanta University; Mahmoud Soliman, MD, Study Chair — Cairo University; Waleed Tawfeek, MD, Study Chair — Benha University; Ahmed Saber, MD, Study Chair — Benha University; Amr Abdelrahman, Study Chair — Zagazig University
Locations (1):
- Ayman Shehata Dawood, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We will decide the type of data to share
Supporting Information: Study Protocol
Time Frame: 3 months